CLINICAL TRIAL: NCT03286998
Title: The Efficacy of Ultrasound in Predicting Operative Findings and Co-morbidities in Cesarean Section Among Cases of Placenta Accreta
Brief Title: Ultrasound in Prediction of Operative Findings in Cesarean Section Among Placenta Accreta Cases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, assistant professor of obstetrics and gynecology, Cairo University
Other Study IDs: 110149
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Placenta Accreta; Placenta Previa
Keywords: placenta previa; color doppler; placenta accreta; ultrasonography
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- placenta previa: pregnant women with singleton living healthy fetus diagnosed as having placenta previa by grey scale ultrasound (placental tissue covers the internal cervical os or within 2 cm from it)

SUMMARY:
A total of 60 women pregnant more than 28 weeks gestation will be recruited from obstetric outpatient clinic (faculty of medicine -Cairo University Hospital) after being diagnosed of having placenta previa or low lying placenta by grey scale ultrasound. Placenta will be reexamined by grey scale ultrasound & color Doppler. Sonographic parameters evaluated will include placental location, loss of retro-placental clear zone, irregularity and thickness of the uterine-placental interface, the smallest myometrial thickness in sagittal and transverse planes, presence of lacunar spaces and bridging vessels & the presence of abnormal vasculature. The sonographic findings will be compared with intraoperative ones. Hysterectomy specimen (if any was done) will be evaluated histo-pathologically to assess the degree of placental invasion & to confirm the accreta status. The aim of the study is to determine the efficacy of ultrasound in predicting operative findings and associated co-morbidties among cases of placenta accreta.

DETAILED DESCRIPTION:
60 pregnant women with singleton living healthy fetus diagnosed as having placenta previa by grey scale ultrasound and candidate for repeated elective cesarean section (CS) or elective cesarean hysterectomy (if the diagnosis of placenta accreta is confirmed) will be included in the study. Inclusion criteria include: maternal age between 20 & 40 years old, gestational age more than 28 weeks (confirmed by a reliable date for the last menstrual period and 1st trimester ultrasound scan), one or more cesarean section scar & the presence of placenta previa with high possibility of being placenta accreta when scanned by grey scale ultrasound. Women who had chronic or pregnancy induced diseases or any emergency or unplanned CS will be excluded. Informed consents will be obtained from all patients after explanation of the aim of the study & the potential risks. For all patients, full history will be taken followed by complete physical examination & routine obstetric ultrasound (to confirm the presence of placenta previa i.e. placental tissue covers the internal cervical os or within 2 cm from it). For all Participants, the placentae will be reexamined in systematic manner by gray-scale & color Doppler ultrasound via transabdominal and/or transvaginal approach using Volusion Pro-V ultrasonography machine (GE Healthcare Austria GmbH, Seoul, Korea). All exams will be done by expert sonographer & the possibility of concomitant placenta accreta will be checked. The placenta will be scanned with adequate bladder volume to visualize the bladder- uterine serosal interface correctly & the angle of insonation will kept as low as possible. The presence of one or more of the following features in grey scale ultrasound will be indicative of placenta accreta (presence of abnormal placental lacunae / complete loss of retroplacental sonolucent zone / myometrial thinning / disruption of the uterine serosa-bladder interface / presence of mass invading the urinary bladder). Similarly, placenta accreta will be diagnosed by the presence of at least one of the following features in color Doppler scan: diffuse or focal lacunar flow - sonolucent vascular lakes - hypervascularity of the utero-vesical interface with bridging vessels connecting the placenta to the bladder). The sonographic provisional diagnosis (i.e placenta previa, focal accreta, accreta , increta or percreta) with the concomitant invasion of adjacent structures (e.g., the urinary bladder) will be documented. For all participants, termination of pregnancy will be by elective CS or elective cesarean hysterectomy. Furthermore, operative findings as regard the placenta and the invasion of adjacent structures will be documented. All operative procedures will be done by senior staff obstetrician with special interest in placenta accreta. For hysterectomy specimens, histopathological examination will be done to assess the degree of myometrial invasion & to confirm the diagnosis of placenta accreta. Maternal morbidities (i.e. massive bleeding with the need of blood transfusion, pelvic organ injury or ICU admission) or mortalities will be documented. Neonatal morbidities (i.e. prematurity or NICU admission) or mortalities will be documented. The ultrasonographic findings will be compared to operative details and histopathological reports. The aim of the study is to evaluate the efficacy of ultrasound in predicting operative findings and associated co-morbidities among cases of placenta accreta.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 20 & 40 years old
* Singleton living healthy fetus.
* Having placenta previa by grey scale ultrasound with high possibility of being placenta accreta when scanned by grey scale ultrasound
* Gestational age more than 28 weeks (confirmed by a reliable date for the last menstrual period and 1st trimester ultrasound scan).
* One or more cesarean section scar

Exclusion Criteria:

* Women who had chronic or pregnancy induced diseases
* Emergency or unplanned CS will be performed.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 60 women pregnant more than 28 weeks gestation will be recruited from obstetric outpatient clinic (faculty of medicine -Cairo University Hospital) after being diagnosed of having placenta previa or low lying placenta by grey scale ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
the accuracy of ultrasound in predicting operative finding in cases of placenta accreta | during cesarean section or elective cesarean hysterectomy
  compare ultrasound report findings with the operative details report in hospital records

CONTACTS AND LOCATIONS:
Overall Officials: Moutaz Elsherbini, M.D, Principal Investigator — Assistant professor of obstetrics and gynecology - Cairo university
Locations (2):
- Egypt (2):
  - Kasr Elainy Hospital (Cairo University), Cairo
  - Faculty of medicine- Cairo university, Cairo